CLINICAL TRIAL: NCT00225654
Title: The ELUTES Clinical Trial (European Evaluation of Paclitaxel Eluting Stent)
Brief Title: The ELUTES Clinical Trial
Acronym: ELUTES I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 505
Record Dates: First submitted 2005-09-12; First posted 2005-09-26 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery; stent; drug eluting; patency; restenosis
MeSH Terms: conditions — Coronary Artery Disease

INTERVENTIONS:
Device: coronary stent

SUMMARY:
ELUTES is a European multicenter, randomized, controlled, triple-blinded study designed to evaluate the ability of the Paclitaxel Eluting V-Flex Plus coronary stent to reduce restenosis in the coronary artery.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be eligible to undergo planned treatment of a single de novo lesion in a native coronary artery.
* Patient must be an acceptable candidate for coronary artery bypass surgery.
* Patient or legal guardian must have signed informed consent.
* Patient agrees to return at one month for an office visit to assess cardiovascular status and at 6 months for an office visit to assess cardiovascular status and for a diagnostic angiogram.

Exclusion Criteria:

* Patient must be less than 18 years old.
* Patient has history of bleeding diathesis or coagulopathy or will refuse blood transfusions.
* Patient is simultaneously participating in another investigative interventional cardiovascular device or drug study.
* Patient has known hypersensitivity or contraindication to aspirin, clopidogrel, or stainless steel, or a sensitivity to contrast dye.
* Women of child bearing potential.
* Patient has other medical condition that may cause non-compliance with the protocol, confound the results, or is associated with limited life expectancy.
* Patient has been diagnosed with a myocardial infarction within 72 hours prior to procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192
Dates: Start 2000-01; Study Completion 2001-11

PRIMARY OUTCOMES:
Angiographic in-stent % diameter stenosis and late loss at follow up.

SECONDARY OUTCOMES:
Major adverse events
Total lesion revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Gershlick, MD, Principal Investigator — Glenfield Hospital
Locations (1):
- Contact Sponsor, Bloomington, Indiana, United States